CLINICAL TRIAL: NCT04996264
Title: Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of a Multi-Dose Regimen of Oral Varespladib-Methyl in Subjects Bitten by Venomous Snakes
Brief Title: Broad-spectrum Rapid Antidote: Varespladib Oral for Snakebite
Acronym: BRAVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophirex, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPX-PR-01
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Snakebites; Envenoming; Envenoming, Snake; Envenomation, Snake
Keywords: envenoming; venom; snakebite; snakebite severity score; varespladib; snake; antidote; LY333013; sPLA2
MeSH Terms: conditions — Snake Bites | interventions — varespladib methyl; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, Investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment except for a specified unblinded statistician and programmer from the study contract research organization who will have access to the randomization code. The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data to all study-related personnel upon database lock. If an interim analysis is conducted, then unblinded personnel who are not otherwise involved in the study will prepare the data for review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varespladib-methyl (Experimental): Varespladib-methyl is an immediate-release (IR), oval, white, film-coated tablet at a dosage strength of 250 mg for oral administration.
  Scaled pediatric doses of varespladib-methyl are supplied as 50 mg IR capsules for oral administration.
  Adult subjects will receive an initial loading dose of 500 mg (2 × 250 mg oral tablet) varespladib-methyl upon randomization, followed by dosing with 250 mg varespladib-methyl (1 × 250 mg oral tablet) approximately 12 hours later, and subsequent twice daily (BID) dosing with 1 × 250 mg varespladib-methyl oral tablets for the remainder of the 7-day treatment period. Tablets may be administered via naso- or orogastric tubes in patients requiring mechanical ventilation.
  Pediatric subjects (5 to < 18 years) will be administered doses of varespladib-methyl determined by allometric scaling, provided as 50 mg capsules. Age-appropriate capsules may be administered via naso- or orogastric tubes in patients requiring mechanical ventilation.
  Interventions: Drug: Varespladib Methyl; Drug: Standard of care (SOC)
- Placebo (Placebo Comparator): The oral placebo is supplied as a white film-coated oval tablet to match the appearance of the varespladib-methyl 250 mg tablet and contains a subset of the excipients present in the active tablet formulation: lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Placebo for scaled pediatric dosing is supplied as an immediate-release capsule to match the varespladib-methyl 50 mg capsule, and contains the excipients lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  The dosing of placebo will match that of varespladib-methyl.
  Interventions: Drug: Placebo; Drug: Standard of care (SOC)

INTERVENTIONS:
Drug: Varespladib Methyl — Varespladib-methyl (LY333013) is an IR, oval, white, film-coated tablet at a dosage strength of 250 mg for oral administration. Scaled pediatric doses of varespladib-methyl (LY333013) are supplied as 50 mg IR capsules for oral administration.
  Other Names: LY333013
  Arms: Varespladib-methyl
Drug: Placebo — The oral placebo is supplied as a white film-coated oval tablet to match the appearance of the varespladib-methyl 250 mg tablet and contains a subset of the excipients present in the active tablet formulation: lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Placebo for scaled pediatric dosing is supplied as an IR capsule to match the varespladib-methyl 50 mg capsule, and contains the excipients lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Arms: Placebo
Drug: Standard of care (SOC) — SOC (including antivenom) will continue to be administered throughout the subject's participation in the study according to the protocol and the judgment of the Investigator.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, phase 2 study designed to evaluate the safety, tolerability and efficacy of varespladib-methyl, concurrently with standard of care (SOC), in subjects bitten by venomous snakes.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, phase 2 study designed to evaluate the safety, tolerability, and efficacy of varespladib-methyl, concurrently with SOC, in subjects bitten by venomous snakes.

Approximately 110 male and female eligible subjects will be enrolled and randomized to receive active varespladib-methyl or placebo (in addition to SOC) in a 1:1 ratio (approximately 36 per group). There will be no stratification by type of snakebite, though randomization will be stratified by age group (5 to 11 years, 12 to 17 years, and ≥ 18 years) and by the presence or absence of severe neurologic symptoms defined by yes/no neurologic system subscore of the snakebite severity score of ≥ 2.

Effective treatments for snakebite envenoming represents a deadly and unmet global medical need. While antivenoms comprise the SOC for treatment of snakebites, they suffer from several limitations including specificity of each antivenom for specific species of snake, limited access to antivenom in rural areas, practical storage requirements, and delays in administration. Treatment of snakebite envenoming with the small-molecule drug varespladib-methyl, which targets secreted phospholipase A₂ (sPLA₂) present in more than 95% of snake venoms, has the potential to overcome several limitations of serum-based antivenoms that underpin traditional SOC.

This study in the United States and India will provide coverage of a broad spectrum of venomous snake genera, including elapids, pit vipers, and potentially exotics such as vipers and colubrids if encountered over the course of the study. The study is designed to cover differing geographies and differing sPLA₂ structures. Study sites have been and will be selected based on demonstrated historical incidence of snake bites from species deemed relevant to this study, to ensure a broad range of envenoming toxins are expected to be encountered in potential study subjects.

The study design allows for both treatment arms (varespladib-methyl and placebo) to receive SOC (e.g., antivenom) concurrently. Thus, critically ill adult and pediatric subjects may receive emergency treatment in a timely manner while being evaluated for the potential clinical benefit associated with inhibition of venom sPLA₂ and inflammatory sPLA2s by varespladib-methyl.

Because subjects with severe snakebites are admitted to emergency departments, this study was designed to screen, enroll, and administer treatment in a single visit at the hospital upon admission. Because varespladib-methyl is administered orally, subjects who demonstrate substantial improvement and are eligible for discharge from the hospital may continue investigational product treatment in an outpatient setting.

Risks associated with the control (placebo) arm of this study include the same risks associated with SOC (antivenom).

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female subject ≥ 5 years of age with venomous snakebite and must present with an initial SSS of

   * 2 points in any SSS category other than gastrointestinal and 1 or more additional points in any other SSS category other than gastrointestinal or
   * ≥ 3 in any SSS category other than gastrointestinal.

   SSS scoring should be performed for inclusion assessment without waiting for receipt of Baseline hematological laboratory results. Gastrointestinal scores should not be used for inclusion.
2. Index event (snakebite) must be symptomatic and must have occurred within 10 hours of eligibility assessment.
3. Must meet one of two categories of inclusion criteria:

   Category 1: The patient has not yet completed first dose of antivenom:

   SSS inclusion score* of ≥2 in one system and ≥1 in another system (2+1) OR ≥3 in at least one system.

   OR

   Category 2: The patient has completed an initial dose of antivenom:

   SSS inclusion score* of ≥2 in one system and ≥1 in another system (2+1) OR ≥3 in at least one system AND CGI-I score of ≥5 (i.e., minimally worse, much worse, or very much worse).
4. Is willing (or legally authorized representative is willing) to provide informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Has received antivenom treatment for envenoming prior to enrollment in this study.
2. Is considered by the investigator to have a clinically significant upper GI bleed evidenced by hematemesis, "coffee-ground" emesis or nasogastric aspirate, or hematochezia thought to originate from upper GI tract.
3. Has history of cerebrovascular accident or intracranial bleeding of any kind, acute coronary syndrome, myocardial infarction, or severe pulmonary hypertension.
4. Has known history of inherited bleeding or coagulation disorder.
5. Is, at Screening Visit, using the following anticoagulants: warfarin/coumadin, argatroban, bivalirudin, lepirudin, apixaban, dabigatran, clopidogrel, prasugrel, ticlopidine or another anticoagulant agent not specifically listed, or has used heparin, enoxaparin, fondaparinux, or other low molecular weight heparin or antiarrhythmic drugs within 14 days prior to treatment.
6. Has a history of chronic liver disease such as chronic active viral hepatitis, alcohol-related liver disease, non-alcoholic steatohepatitis, non-alcoholic fatty liver disease, hemochromatosis, primary biliary cirrhosis, primary sclerosing cholangitis, or autoimmune hepatitis.
7. Reports or has known pre-existing renal impairment or chronic kidney disease (defined as Stage 4 or receiving dialysis or hemofiltration).
8. Has a known allergy or significant adverse reaction to varespladib-methyl or related compounds.
9. Is considered by the Investigator to be unable to comply with protocol requirements due to geographic considerations, psychiatric disorders, or other compliance concerns.
10. Is pregnant, has a positive serum human chorionic gonadotropin (hCG) pregnancy test or not willing to use a highly effective method of contraception for 14 days after initial treatment, or is breast-feeding.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lewin, MD, PhD, Principal Investigator — Ophirex, Inc.; Timothy F Platts-Mills, MD, MSc, Principal Investigator — Ophirex, Inc.
Locations (16):
- United States (8):
  - University of Arizona, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Florida Health, Jacksonville, Florida
  - Agusta University Medical Center, Augusta, Georgia
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - LSU LA Poison Control Center, Shreveport, Louisiana
  - University of Mississippi Medical Center - Jackson, Jackson, Mississippi
  - Duke University Hospital Durham, NC, Durham, North Carolina
- India (8):
  - Government medical College, Kozhikode, Calicut
  - Father Muller medical College Hospital, Mangalore, Karnataka
  - K R Hospital Mysore medical College and Research Institute, Mysore, Karnataka
  - Jubilee Mission Medical College and Research Institute, Thrissur, Kerala
  - Jawaharlal Institute of Postgraduate Medical Education & Research, Puducherry, Puducherry
  - S.P. Medical College Snakebite Research Cell, Bikaner, Rajasthan
  - Calcutta National Medical College, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varespladib. Am J Cardiovasc Drugs. 2011;11(2):137-43. doi: 10.2165/11533650-000000000-00000. PMID 21446779
- [Background] Alangode A, Rajan K, Nair BG. Snake antivenom: Challenges and alternate approaches. Biochem Pharmacol. 2020 Nov;181:114135. doi: 10.1016/j.bcp.2020.114135. Epub 2020 Jul 3. PMID 32628928
- [Background] Albulescu LO, Xie C, Ainsworth S, Alsolaiss J, Crittenden E, Dawson CA, Softley R, Bartlett KE, Harrison RA, Kool J, Casewell NR. A therapeutic combination of two small molecule toxin inhibitors provides broad preclinical efficacy against viper snakebite. Nat Commun. 2020 Dec 15;11(1):6094. doi: 10.1038/s41467-020-19981-6. PMID 33323937
- [Background] Anderson BO, Moore EE, Banerjee A. Phospholipase A2 regulates critical inflammatory mediators of multiple organ failure. J Surg Res. 1994 Feb;56(2):199-205. doi: 10.1006/jsre.1994.1032. PMID 8121178
- [Background] Arce-Bejarano R, Lomonte B, Gutierrez JM. Intravascular hemolysis induced by the venom of the Eastern coral snake, Micrurus fulvius, in a mouse model: identification of directly hemolytic phospholipases A2. Toxicon. 2014 Nov;90:26-35. doi: 10.1016/j.toxicon.2014.07.010. Epub 2014 Aug 1. PMID 25088177
- [Background] Bittenbinder MA, Zdenek CN, Op den Brouw B, Youngman NJ, Dobson JS, Naude A, Vonk FJ, Fry BG. Coagulotoxic Cobras: Clinical Implications of Strong Anticoagulant Actions of African Spitting Naja Venoms That Are Not Neutralised by Antivenom but Are by LY315920 (Varespladib). Toxins (Basel). 2018 Dec 4;10(12):516. doi: 10.3390/toxins10120516. PMID 30518149
- [Background] Bryan-Quiros W, Fernandez J, Gutierrez JM, Lewin MR, Lomonte B. Neutralizing properties of LY315920 toward snake venom group I and II myotoxic phospholipases A2. Toxicon. 2019 Jan;157:1-7. doi: 10.1016/j.toxicon.2018.11.292. Epub 2018 Nov 14. PMID 30447275
- [Background] Bulfone TC, Samuel SP, Bickler PE, Lewin MR. Developing Small Molecule Therapeutics for the Initial and Adjunctive Treatment of Snakebite. J Trop Med. 2018 Jul 30;2018:4320175. doi: 10.1155/2018/4320175. eCollection 2018. PMID 30154870
- [Background] Chippaux JP. Estimate of the burden of snakebites in sub-Saharan Africa: a meta-analytic approach. Toxicon. 2011 Mar 15;57(4):586-99. doi: 10.1016/j.toxicon.2010.12.022. Epub 2011 Jan 9. PMID 21223975
- [Background] Fernandez ML, Quartino PY, Arce-Bejarano R, Fernandez J, Camacho LF, Gutierrez JM, Kuemmel D, Fidelio G, Lomonte B. Intravascular hemolysis induced by phospholipases A2 from the venom of the Eastern coral snake, Micrurus fulvius: Functional profiles of hemolytic and non-hemolytic isoforms. Toxicol Lett. 2018 Apr;286:39-47. doi: 10.1016/j.toxlet.2017.11.037. Epub 2017 Nov 29. PMID 29197624
- [Background] Fontana Oliveira IC, Gutierrez JM, Lewin MR, Oshima-Franco Y. Varespladib (LY315920) inhibits neuromuscular blockade induced by Oxyuranus scutellatus venom in a nerve-muscle preparation. Toxicon. 2020 Nov;187:101-104. doi: 10.1016/j.toxicon.2020.08.023. Epub 2020 Sep 2. PMID 32889027
- [Background] Gerardo CJ, Vissoci JRN, Evans CS, Simel DL, Lavonas EJ. Does This Patient Have a Severe Snake Envenomation?: The Rational Clinical Examination Systematic Review. JAMA Surg. 2019 Apr 1;154(4):346-354. doi: 10.1001/jamasurg.2018.5069. PMID 30758508
- [Background] Gutierrez JM, Calvete JJ, Habib AG, Harrison RA, Williams DJ, Warrell DA. Snakebite envenoming. Nat Rev Dis Primers. 2017 Sep 14;3:17063. doi: 10.1038/nrdp.2017.63. PMID 28905944
- [Background] Gutierrez JM, Lewin MR, Williams DJ, Lomonte B. Varespladib (LY315920) and Methyl Varespladib (LY333013) Abrogate or Delay Lethality Induced by Presynaptically Acting Neurotoxic Snake Venoms. Toxins (Basel). 2020 Feb 20;12(2):131. doi: 10.3390/toxins12020131. PMID 32093386
- [Background] Halilu S, Iliyasu G, Hamza M, Chippaux JP, Kuznik A, Habib AG. Snakebite burden in Sub-Saharan Africa: estimates from 41 countries. Toxicon. 2019 Mar 1;159:1-4. doi: 10.1016/j.toxicon.2018.12.002. Epub 2018 Dec 27. PMID 30594637
- [Background] Kazandjian TD, Petras D, Robinson SD, van Thiel J, Greene HW, Arbuckle K, Barlow A, Carter DA, Wouters RM, Whiteley G, Wagstaff SC, Arias AS, Albulescu LO, Plettenberg Laing A, Hall C, Heap A, Penrhyn-Lowe S, McCabe CV, Ainsworth S, da Silva RR, Dorrestein PC, Richardson MK, Gutierrez JM, Calvete JJ, Harrison RA, Vetter I, Undheim EAB, Wuster W, Casewell NR. Convergent evolution of pain-inducing defensive venom components in spitting cobras. Science. 2021 Jan 22;371(6527):386-390. doi: 10.1126/science.abb9303. PMID 33479150
- [Background] Le Geyt J, Pach S, Gutierrez JM, Habib AG, Maduwage KP, Hardcastle TC, Hernandez Diaz R, Avila-Aguero ML, Ya KT, Williams D, Halbert J. Paediatric snakebite envenoming: recognition and management of cases. Arch Dis Child. 2021 Jan;106(1):14-19. doi: 10.1136/archdischild-2020-319428. Epub 2020 Oct 28. PMID 33115713
- [Background] Lewin M, Samuel S, Merkel J, Bickler P. Varespladib (LY315920) Appears to Be a Potent, Broad-Spectrum, Inhibitor of Snake Venom Phospholipase A2 and a Possible Pre-Referral Treatment for Envenomation. Toxins (Basel). 2016 Aug 25;8(9):248. doi: 10.3390/toxins8090248. PMID 27571102
- [Background] Lewin MR, Gilliam LL, Gilliam J, Samuel SP, Bulfone TC, Bickler PE, Gutierrez JM. Delayed LY333013 (Oral) and LY315920 (Intravenous) Reverse Severe Neurotoxicity and Rescue Juvenile Pigs from Lethal Doses of Micrurus fulvius (Eastern Coral Snake) Venom. Toxins (Basel). 2018 Nov 17;10(11):479. doi: 10.3390/toxins10110479. PMID 30453607
- [Background] Lewin MR, Gutierrez JM, Samuel SP, Herrera M, Bryan-Quiros W, Lomonte B, Bickler PE, Bulfone TC, Williams DJ. Delayed Oral LY333013 Rescues Mice from Highly Neurotoxic, Lethal Doses of Papuan Taipan (Oxyuranus scutellatus) Venom. Toxins (Basel). 2018 Sep 20;10(10):380. doi: 10.3390/toxins10100380. PMID 30241297
- [Background] Longbottom J, Shearer FM, Devine M, Alcoba G, Chappuis F, Weiss DJ, Ray SE, Ray N, Warrell DA, Ruiz de Castaneda R, Williams DJ, Hay SI, Pigott DM. Vulnerability to snakebite envenoming: a global mapping of hotspots. Lancet. 2018 Aug 25;392(10148):673-684. doi: 10.1016/S0140-6736(18)31224-8. Epub 2018 Jul 17. PMID 30017551
- [Background] Pach S, Le Geyt J, Gutierrez JM, Williams D, Maduwage KP, Habib AG, Gustin R, Avila-Aguero ML, Ya KT, Halbert J. Paediatric snakebite envenoming: the world's most neglected 'Neglected Tropical Disease'? Arch Dis Child. 2020 Dec;105(12):1135-1139. doi: 10.1136/archdischild-2020-319417. Epub 2020 Sep 30. PMID 32998874
- [Background] PARRISH HM. SNAKE VENENATION IN ILLINOIS. IMJ Ill Med J. 1965 Jun;127:671-7. No abstract available. PMID 14295634
- [Background] Prasarnpun S, Walsh J, Awad SS, Harris JB. Envenoming bites by kraits: the biological basis of treatment-resistant neuromuscular paralysis. Brain. 2005 Dec;128(Pt 12):2987-96. doi: 10.1093/brain/awh642. Epub 2005 Sep 29. PMID 16195243
- [Background] Ruha AM, Kleinschmidt KC, Greene S, Spyres MB, Brent J, Wax P, Padilla-Jones A, Campleman S; ToxIC Snakebite Study Group. The Epidemiology, Clinical Course, and Management of Snakebites in the North American Snakebite Registry. J Med Toxicol. 2017 Dec;13(4):309-320. doi: 10.1007/s13181-017-0633-5. Epub 2017 Oct 3. PMID 28975491
- [Background] Salvador GHM, Gomes AAS, Bryan-Quiros W, Fernandez J, Lewin MR, Gutierrez JM, Lomonte B, Fontes MRM. Structural basis for phospholipase A2-like toxin inhibition by the synthetic compound Varespladib (LY315920). Sci Rep. 2019 Nov 20;9(1):17203. doi: 10.1038/s41598-019-53755-5. PMID 31748642
- [Background] Sankar J, Nabeel R, Sankar MJ, Priyambada L, Mahadevan S. Factors affecting outcome in children with snake envenomation: a prospective observational study. Arch Dis Child. 2013 Aug;98(8):596-601. doi: 10.1136/archdischild-2012-303025. Epub 2013 May 28. PMID 23716133
- [Background] Schulte J, Domanski K, Smith EA, Menendez A, Kleinschmidt KC, Roth BA. Childhood Victims of Snakebites: 2000-2013. Pediatrics. 2016 Nov;138(5):e20160491. doi: 10.1542/peds.2016-0491. PMID 27940763
- [Background] Seifert SA, Boyer LV, Benson BE, Rogers JJ. AAPCC database characterization of native U.S. venomous snake exposures, 2001-2005. Clin Toxicol (Phila). 2009 Apr;47(4):327-35. doi: 10.1080/15563650902870277. PMID 19514880
- [Background] Snyder DW, Bach NJ, Dillard RD, Draheim SE, Carlson DG, Fox N, Roehm NW, Armstrong CT, Chang CH, Hartley LW, Johnson LM, Roman CR, Smith AC, Song M, Fleisch JH. Pharmacology of LY315920/S-5920, [[3-(aminooxoacetyl)-2-ethyl-1- (phenylmethyl)-1H-indol-4-yl]oxy] acetate, a potent and selective secretory phospholipase A2 inhibitor: A new class of anti-inflammatory drugs, SPI. J Pharmacol Exp Ther. 1999 Mar;288(3):1117-24. PMID 10027849
- [Background] Sorensen J, Kald B, Tagesson C, Lindahl M. Platelet-activating factor and phospholipase A2 in patients with septic shock and trauma. Intensive Care Med. 1994 Nov;20(8):555-61. doi: 10.1007/BF01705721. PMID 7706567
- [Background] Tasoulis T, Isbister GK. A Review and Database of Snake Venom Proteomes. Toxins (Basel). 2017 Sep 18;9(9):290. doi: 10.3390/toxins9090290. PMID 28927001
- [Background] Uhl W, Beger HG, Hoffmann G, Hanisch E, Schild A, Waydhas C, Entholzner E, Muller K, Kellermann W, Vogeser M, et al. A multicenter study of phospholipase A2 in patients in intensive care units. J Am Coll Surg. 1995 Mar;180(3):323-31. PMID 7874343
- [Background] Vaiyapuri S, Vaiyapuri R, Ashokan R, Ramasamy K, Nattamaisundar K, Jeyaraj A, Chandran V, Gajjeraman P, Baksh MF, Gibbins JM, Hutchinson EG. Snakebite and its socio-economic impact on the rural population of Tamil Nadu, India. PLoS One. 2013 Nov 21;8(11):e80090. doi: 10.1371/journal.pone.0080090. eCollection 2013. PMID 24278244
- [Background] Williams DJ, Faiz MA, Abela-Ridder B, Ainsworth S, Bulfone TC, Nickerson AD, Habib AG, Junghanss T, Fan HW, Turner M, Harrison RA, Warrell DA. Strategy for a globally coordinated response to a priority neglected tropical disease: Snakebite envenoming. PLoS Negl Trop Dis. 2019 Feb 21;13(2):e0007059. doi: 10.1371/journal.pntd.0007059. eCollection 2019 Feb. No abstract available. PMID 30789906
- [Background] Xie C, Albulescu LO, Bittenbinder MA, Somsen GW, Vonk FJ, Casewell NR, Kool J. Neutralizing Effects of Small Molecule Inhibitors and Metal Chelators on Coagulopathic Viperinae Snake Venom Toxins. Biomedicines. 2020 Aug 20;8(9):297. doi: 10.3390/biomedicines8090297. PMID 32825484
- [Background] Zinenko O, Tovstukha I, Korniyenko Y. PLA2 Inhibitor Varespladib as an Alternative to the Antivenom Treatment for Bites from Nikolsky's Viper Vipera berus nikolskii. Toxins (Basel). 2020 May 29;12(6):356. doi: 10.3390/toxins12060356. PMID 32485836
- See also: Drug Development and Drug Interactions | Table of Substrates, Inhibitors and Inducers — https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers

RESULTS

PARTICIPANT FLOW:
Groups:
- Varespladib-methyl: Varespladib-methyl is an immediate-release (IR), oval, white, film-coated tablet at a dosage strength of 250 mg for oral administration.
  Scaled pediatric doses of varespladib-methyl are supplied as 50 mg IR capsules for oral administration.
  Adult subjects will receive an initial loading dose of 500 mg (2 × 250 mg oral tablet) varespladib-methyl upon randomization, followed by dosing with 250 mg varespladib-methyl (1 × 250 mg oral tablet) approximately 12 hours later, and subsequent twice daily (BID) dosing with 1 × 250 mg varespladib-methyl oral tablets for the remainder of the 7-day treatment period. Tablets may be administered via naso- or orogastric tubes in patients requiring mechanical ventilation.
  Pediatric subjects (5 to < 18 years) will be administered doses of varespladib-methyl determined by allometric scaling, provided as 50 mg capsules. Age-appropriate capsules may be administered via naso- or orogastric tubes in patients requiring mechanical ventilation.
  Varespladib Methyl: Varespladib-methyl (LY333013) is an IR, oval, white, film-coated tablet at a dosage strength of 250 mg for oral administration. Scaled pediatric doses of varespladib-methyl (LY333013) are supplied as 50 mg IR capsules for oral administration.
  Standard of care (SOC): SOC (including antivenom) will continue to be administered throughout the subject's participation in the study according to the protocol and the judgment of the Investigator.
- Placebo: The oral placebo is supplied as a white film-coated oval tablet to match the appearance of the varespladib-methyl 250 mg tablet and contains a subset of the excipients present in the active tablet formulation: lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Placebo for scaled pediatric dosing is supplied as an immediate-release capsule to match the varespladib-methyl 50 mg capsule, and contains the excipients lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  The dosing of placebo will match that of varespladib-methyl.
  Placebo: The oral placebo is supplied as a white film-coated oval tablet to match the appearance of the varespladib-methyl 250 mg tablet and contains a subset of the excipients present in the active tablet formulation: lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Placebo for scaled pediatric dosing is supplied as an IR capsule to match the varespladib-methyl 50 mg capsule, and contains the excipients lactose monohydrate, microcrystalline cellulose, and magnesium stearate.
  Standard of care (SOC): SOC (including antivenom) will continue to be administered throughout the subject's participation in the study according to the protocol and the judgment of the Investigator.
Period: Overall Study
Arm/Group | Varespladib-methyl | Placebo
Started | 45 | 50
Completed | 41 | 43
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — 1 left AMA | 0 | 1
Not completed — Subject changed hospitals | 0 | 1
Not completed — unable to complete due to work | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varespladib-methyl | Placebo | Total
Number analyzed (Participants) | 45 | 50 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 33 | 43 | 76
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (18.6) | 41.9 (15.9) | 39.9 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 35 | 39 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 41 | 47 | 88
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 17 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33
  India | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in the Combined Pulmonary, Cardiovascular, Hematologic, Nervous System, and Renal Subscores of the Snakebite Severity Score (SSS)
Description: Change from baseline (pre-dosing) to 6 and 9 hours after the first dose, in the combined pulmonary, cardiovascular, hematologic symptoms, nervous system, and renal subscores of the SSS. The values from each of these subscores will be totaled. The average of the 6- and 9-hour scores will be used as the post-treatment value.
  The Snakebite Severity Scale (SSS) is a tool used to measure the severity of envenoming based on up to 7 body categories: pulmonary, cardiovascular, gastrointestinal, nervous, and renal system (graded at levels from Grade 0 to Grade 3), local wound, and hematological, (graded at levels from Grade 0 to Grade 4). A higher score indicates worse symptoms. The minimum score for the five item SSS is 0 and the maximum score is 16, with the higher score indicating worse symptoms. For the primary outcome we are focusing only on 5 subscores, that does not include the local wound nor the gastrointestinal subscores.
Time Frame: Baseline to 6 and 9 hours after first dose
Measure: Mean (Standard Error); unit: Snakebite Severity Score
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 50
Snakebite Severity Score | 1.1 (0.3) | 1.5 (0.2)

2. Secondary Outcome: Area Under the Curve (AUC) of the Local Wound, Pulmonary, Cardiovascular, Hematologic Symptoms, Renal, and Nervous System Sections of the SSS
Description: Baseline (pre-dosing) through Day 7 in the AUC of the local wound, pulmonary, cardiovascular, hematologic symptoms, nervous, and renal system sections of the SSS.
  The Snakebite Severity Scale (SSS) is a tool used to measure the severity of envenoming based on 7 body categories: pulmonary, cardiovascular, gastrointestinal, nervous, and renal effects (graded at levels from Grade 0 to Grade 3), local wound and hematological, (graded at levels from Grade 0 to Grade 4). A higher score indicates worse symptoms. The maximum score for the SSS is 23.
  For this outcome, the maximum score is 20 and if this score was present for the entire first week (168 hours) the maximum AUC is 3,370. The minimum AUC is a score of 3 at baseline and a score of 0 at three hours, which gives an AUC of 5.25.
Time Frame: Baseline through Day 7
Measure: Mean (Standard Error); unit: Snakebite severity score X hours
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 50
Snakebite severity score X hours | 421 (45) | 430 (44)

3. Secondary Outcome: Area Under the Curve (AUC) of the Numeric Pain Rating Scale (NPRS)
Description: Numeric Pain Rating Scale is a scale that goes from 0 to 10 with 10 being the worst possible pain. This measure is an AUC measure that is calculated from 0 to 48 hours using trapezoidal function in which the mean score for any given 2 periods of time is multiplied by the elapsed duration of time between those two periods. Each of these mean scores are summed to calculate the AUC. The minimum score is 0 and the maximum is 480.
Time Frame: From Baseline through Day 3
Measure: Mean (Standard Error); unit: scores on a scale * hours
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 50
scores on a scale * hours | 170 (17) | 173 (18)

4. Secondary Outcome: Clinician Global Impression - Improvement
Description: Clinician Global Impression - Improvement focus on improvement for Day 2. The scale is a 1 to 7 score with 1 indicating very much improved and 7 indicating very much worse.
Time Frame: Day 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 50
score on a scale | 2.3 (0.2) | 2.4 (0.2)

5. Secondary Outcome: All-cause Mortality
Description: The number of patients experiencing the event (death). The all-cause mortality will be censored at Day 60.
Time Frame: Baseline through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 50
Participants | 0 | 0

6. Secondary Outcome: Patient-Specific Functional Scale (PSFS) Score
Description: PSFS total score on Day 7. The PSFS is a 3-item instrument which assesses functional abilities. The total score ranges from 0 to 10 with a lower score indicating greater functional difficulties.
Time Frame: Day 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 40 | 41
score on a scale | 5.89 (0.29) | 5.86 (0.29)

7. Secondary Outcome: Numeric Pain Rating Scale (NPRS) Score
Description: Change from baseline (pre-dosing) through Day 28 in NPRS score in patients able to respond pre-dosing through Day 28.
  The Numeric Pain Rating Scale is an 11-point scale for patient self-reporting of pain with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline through Day 28
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 41 | 42
score on a scale | 6.4 (0.2) | 6.1 (0.2)

8. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and AEs Leading to Discontinuation of Investigational Product (IP)
Description: Adverse events will be assessed from the time of signing informed consent to 28 days after initiating study drug.
Time Frame: 28 Days after the initiation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib-methyl | Placebo
Number analyzed (Participants) | 45 | 49
Participants | 19 | 28

ADVERSE EVENTS:
Time Frame: Death was assessed up to 60 days, all other adverse events were assessed up to 28 Days after initiation of study drug.
Arm/Group | Varespladib-methyl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/50
Other Adverse Events (participants affected / at risk) | 19/45 | 28/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varespladib-methyl (N=45) | Placebo (N=50)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Subject experienced hypotensive episode 30 minutes prior to receiving study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varespladib-methyl (N=45) | Placebo (N=50)
headache (Nervous system disorders) | 2 (2) | 5 (5)
Abnormal labs (Blood and lymphatic system disorders) | 7 (9) | 7 (14)
Nausea and vomiting (Gastrointestinal disorders) | 3 (3) | 7 (7)
Infections (Infections and infestations) | 2 (2) | 5 (6)
Anemia and Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT04996264/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT04996264/SAP_001.pdf